CLINICAL TRIAL: NCT06615726
Title: Regular Physical Exercise in Patients With Symptomatic Intracranial Arterial Stenosis: a Prospective Randomized Open-label Blinded Endpoint Trial
Brief Title: Regular Physical Exercise in Patients With Symptomatic Intracranial Arterial Stenosis
Acronym: RESIST
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SPORTS1101
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: Ischemic stroke; Transient Ischemic Attack; Symptomatic intracranial arterial stenosis
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular physical exercise group (Experimental)
  Interventions: Behavioral: Regular physical exercise
- Control group (Other)
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: Regular physical exercise — Best medical treatment plus regular physical exercise. Each subject is equipped with an exercise guidance expert to regularly guide and adjust the exercise plan according to the subject's personal conditions throughout the trial period. After randomization, the exercise guidance expert formulated an individualized aerobic exercise plan based on the subject's preferences and their own exercise abilities. After each exercise, subjects filled out the exercise diary , and reported back to the exercise guidance expert.
  Arms: regular physical exercise group
Other: Control group — Best medical treatment
  Arms: Control group

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of regular physical exercise in preventing ischemic stroke events in patients with symptomatic intracranial arterial stenosis.

DETAILED DESCRIPTION:
The intracranial atherosclerotic stenosis (ICAS) is a common cause of ischemic stroke, and the result of increasing global burden of stroke. There are significant racial differences in the incidence of ICAS, which account for 8%-10% of stroke causes in North America and 30%-50% in Asia. In China, the incidence of ICAS in patients with ischemic stroke or transient ischemic attack (TIA) is as high as 46.6%. Previous studies have shown that stroke patients with ICAS have more severe symptoms, longer hospital stay and higher stroke recurrence rate, and the recurrence rate of stroke increases with the increase of stenosis degree. In the WASID (Warfarin-Aspirin Symptomatic Intracranial Disease trial and several prospective cohort studies) trial, the risk of recurrent stroke remained high even after aggressive medication and risk factor intervention in ICAS patients.

At present, the treatment of ICAS mainly includes drug therapy and endovascular therapy. Both the SAMMPRIS (Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis) trial in 2011 and the VISSIT (the Vitesse Intracranial Stent Study for Ischemic Stroke Therapy) trial in 2015, showed that aggressive medical treatment is more effective and safer than endovascular treatment . A 2018 review comparing stenting versus aggressive medical treatment for symptomatic ICAS also noted that medical treatment remains the preferred treatment for symptomatic ICAS patients compared to endovascular therapy. The results of the CASSISS trial in 2022, showed that endovascular therapy failed to show long-term benefit in severe patients with symptomatic ICAS. However, the above trials also found that even with aggressive medical treatment including dual antiplatelet therapy and intensive management of vascular risk factors, the one-year stroke recurrence rate in patients with symptomatic ICAS is still as high as 20%. This seriously endangers national lives and health, and restricts social and economic development. Therefore, there is an urgent need to explore new treatments to improve patient survival.

Several previous studies have shown that physical exercise can reduce the incidence of all-cause stroke, cardiovascular disease and death, but little is known whether it can reduce the recurrence rate of stroke in patients with symptomatic ICAS. A subgroup analysis of the 2016 SAMMPPRIS trial found that in high-risk symptomatic ICAS patients, physical exercise significantly reduced the likelihood of recurrent stroke, myocardial infarction, or vascular death. A 2023 cross-sectional study that included NOMAS (Northern Manhattan Study) data showed a strong negative association between physical exercise and asymptomatic high-risk ICAS and was not regulated by vascular risk factors. Therefore, this trial conducts a multicenter, randomized, controlled, blinded trial of patients with symptomatic ICAS within 30 days to compare them with a control group that received only secondary stroke prevention health education to determine the association between regular physical exercise and stroke recurrence rates within 1 year in patients with symptomatic ICAS.

ELIGIBILITY:
1. Inclusion criteria:

1. Age ≥40 years and ≤80 years;
2. Ischemic stroke or TIA (transient ischemic attack) onset ≤30 days;
3. Ischemic stroke or TIA is attributed to 50-99% of the ICAS (internal carotid artery, M1 segment of middle cerebral artery, M2 segment of middle cerebral artery, basilar artery, or vertebral artery; the degree of stenosis is determined by magnetic resonance angiography, computed tomography angiography, digital subtraction angiography using the standards of warfarin-aspirin symptomatic intracranial disease );
4. mRS (modified Rankin Scale)≤4;
5. The patient himself or his legal representative signs the informed consent form.

2. Exclusion criteria:

1. Stroke progression within the past 3 days (defined as an increase in the score of National Institute of Health Stroke Scale ≥4 points or an increase in individual items of ≥2 points).
2. mRS≥1 before the stroke onset.
3. Concurrent osteoarthritis, fracture, lower limb venous thrombosis, unstable angina pectoris, respiratory diseases, limb disabilities, etc., making it theoretically difficult to cooperate with the physical activity plan for this trial.
4. Complicated with motor disorders such as Parkinson's disease and Parkinson's syndrome.
5. The vessels responsible for this stroke had tandem lesions (more than 50% of extracranial artery stenosis).
6. The vessel responsible for this stroke has undergone intracranial balloon angioplasty and/or stent implantation (except for mechanical thrombectomy and/or aspiration alone).
7. It is expected that intracranial arterial balloon angioplasty and/or stent implantation will be performed on the vessel responsible for the stroke within 3 months.
8. Patients who exercised regularly within the last 6 months. Regular exercise is defined as four or more moderate intensity exercises per week for more than 10 minutes each time or two or more high intensity exercises per week for more than 10 minutes each time.
9. Inability to understand and/or comply with the trial procedures and/or follow-up due to mental illness, cognitive or emotional disorders.
10. Life expectancy is less than one year.
11. Women who are known to be pregnant or nursing, or have a positive pregnancy test;
12. Are participating in other drug or device research.
13. There are other circumstances that investigators consider are not suitable for enrollment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
New ischemic stroke events | 1 year

SECONDARY OUTCOMES:
New ischemic stroke and transient ischemic attack events in the responsible vessel supply area | 1 year
New ischemic stroke and transient ischemic attack events | 1 year
Hemorrhagic stroke event | 1 year
Myocardial infarction | 1 year
The proportion of modified Rankin Scale score 0-1 (range, 0 to 6, with higher scores indicating greater disability) | 1 year
The score of min montreal cognitive assessment(range, 0 to 15, with higher scores indicating greater cognition) | 1 year
The score of Euro-QoL-5 Dimension(range, 0 to 100, with higher scores indicating better quality of life) | 1 year

OTHER OUTCOMES:
Falls | 1 year
All-cause death | 1 year

CONTACTS AND LOCATIONS:
Locations (58):
- China (58):
  - Taihe Hospital of Traditional Chinese Medicine, Fuyang, Anhui
  - Huainan Sunshine Xinkang Hospital, Huainan, Anhui
  - Suzhou Municipal Hospital, Suzhou, Anhui
  - The Second People's Hospital of Wuhu, Wuhu, Anhui
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Pinggu District Hospital, Beijing, Beijing Municipality
  - Chongqing Sanbo Jiangling Hospital, Chongqing, Chongqing Municipality
  - Zhangzhou Hospital, Zhangzhou, Fu
  - Foshan Fifth People's Hospital, Foshan, Guangdong
  - Foshan Nanhai District Sixth People's Hospital, Foshan, Guangdong
  - Brain Hospital Affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - Longchuan Hospital of Traditional Chinese Medicine, Heyuan, Guangdong
  - Hospital 925, Joint Logistics Support Force, Guizhou, Guiyang
  - Cangzhou People's Hospital of integrated Chinese and Western Medicine, Hebei Province, Cangzhou, Hebei
  - Army Military Medical University Officer School affiliated hospital, Shijiazhuang, Hebei
  - Tangshan Workers' Hospital, Tangshan, Hebei
  - Ningjin County Hospital, Xingtai, Hebei
  - Gongyi Xinhua Hospital of Traditional Chinese Medicine, Gongyi, Henan
  - Tongxu First Hospital, Kaifeng, Henan
  - Fangcheng County People's Hospital, Nanyang, Henan
  - Nanyang City Center Hospital, Nanyang, Henan
  - Shangqiu First People's Hospital, Shangqiu, Henan
  - Yongcheng Central Hospital, Shangqiu, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan
  - Zhengzhou First People's Hospital, Zhengzhou, Henan
  - Zhengzhou Zhongkang Hospital, Zhengzhou, Henan
  - Zhongmou County People's Hospital, Zhengzhou, Henan
  - Xihua County People's Hospital, Zhoukou, Henan
  - Lichuan Ethnic Chinese Medicine Hospital, Lichuan, Hubei
  - Hubei Third People's Hospital, Wuhan, Hubei
  - Yueyang City People's Court, Yueyang, Hubei
  - Liuyang City Jili Hospital, Guankou, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Jiujiang First People's Hospital, Jiujiang, Jiangxi
  - Jilin City People's Hospital, Jilin, Jilin
  - Xinmin People's Hospital, Shenyang, Liaoning
  - Affiliated Hospital of Inner Mongolia University for Nationalities, Tongliao, Neimenggu
  - Yantai Yeda Hospital, Yantai, Shaanxi
  - Shandong University Qilu Hospital Dezhou Hospital, Dezhou, Shandong
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Jinan High-tech East District Hospital, Jinan, Shandong
  - Laixi People's Hospital, Laixi, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Lanshan District People's Hospital, Rizhao, Shandong
  - Affiliated Hospital of Shandong Second Medical University, Weifang, Shandong
  - Yantai Fushan District People's Hospital, Yantai, Shandong
  - Tengzhou Central Hospital, Zaozhuang, Shandong
  - Ningjin County People's Hospital, Dezhou, Shangdong
  - Shanghai Hechuan Rhein Hospital of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Sichuan Academy of Sciences Hospital, Chengdu, Sichuan
  - Jianyang City Hospital of Traditional Chinese Medicine, Jiancheng, Sichuan
  - Ya 'an People's Hospital, Yaan, Sichuan
  - Shihezi People's Hospital, Shihezi, Xinjiang
  - Yongjia County People's Hospital, Wenzhou, Zhejiang
  - Yueqing People's Hospital, Wenzhou, Zhejiang